CLINICAL TRIAL: NCT03503006
Title: Effects of Vitamin D Status on the Outcome of Ivf - Embryo Transfer
Status: Completed | Type: Observational
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Other Study IDs: LCYJ-201802
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2018-03

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At present, there is no agreement on the effect of vitamin D level in serum and follicular fluid on the outcome of IVF-ET pregnancy. Most of these studies were based on the research of total 25 (OH) D, which have ignored that the biological activity of vitamin D molecule is not total 25 (OH) D, but free vitamin D or vitamin D bioavailable, and have flaws in methodology. This project intends to make a prospective cohort study with large sample, based on a complete methodology of total vitamin D and free vitamin D to measure maternal vitamin D levels in blood,to systematically study the effect of maternal vitamin D status on IVF - ET pregnancy outcome. This study is also the first to study the relationship between maternal vitamin D status and the outcome of IVF-ET pregnancy using a complete methodology.

ELIGIBILITY:
Inclusion Criteria:

* female with only fallopian tube factor or male factor infertility,first IVF/ICSI cycle,18 years old≤age≤35 years old,take a long protocol or super-long protocol,18≤BMI≤25, menstrual regularity(periodic change < 7 days)

Exclusion Criteria:

* Hyperprolactinemia, Thyroid dysfunction, uterine malformation ( inadequacy mediastinal uterus ≥1.0cm, Unicornate uterus, double uterus, T Angle of uterus, etc.), uterus adhesion, untreated hydrosalpinx , hysteromyoma（ hysteromyoma≥2.0 cm, and/or Uterine fibroids located within the endometrium≤1cm), endometriosis, diabetes, hypertension, adrenal cortex hyperplasia, Cushing's syndrome, a pituitary amenorrhea

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: the study population will be selected from patients of Reproductive and Genetic Hospital of CITIC-Xiangya
Sampling Method: Non-Probability Sample
Enrollment: 2569 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | Until 28 day after embryo transferred

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China

REFERENCES:
- [Derived] Liu Y, Hocher JG, Ma S, Hu L, Chen H, Zhang X, Gong F, Kramer BK, Lin G, Hocher B. Pre-pregnancy LDL/HDL and total Cholesterol/HDL ratios are strong predictors of gestational diabetes mellitus in women undergoing assisted reproductive technologies. Reprod Biol Endocrinol. 2024 Dec 5;22(1):155. doi: 10.1186/s12958-024-01320-9. PMID 39639281